CLINICAL TRIAL: NCT05113290
Title: Effect and Safety of Recombinant Human Adenovirus Type 5 (H101) in Advanced Hepatocellular Carcinoma Patients With Stable Disease After Sorafenib Treatment: A Randomized, Parallel-Controlled Clinical Trial
Brief Title: Effect and Safety of Recombinant Human Adenovirus Type 5 in Advanced HCC With Stable Disease After Sorafenib Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2021LSK-160
Record Dates: First submitted 2021-10-24; First posted 2021-11-09 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2021-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: oncolytic virus
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- H101+Sorafenib (Experimental): H101 combined with Sorafenib
  Interventions: Drug: Recombinant Human Adenovirus Type 5 injection; Drug: Sorafenib
- Sorafenib (Active Comparator): Patients take Sorafenib only
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Recombinant Human Adenovirus Type 5 injection — Intratumoral injection of lesions with dose of 3 vials (1.5 × 10^12 vp) if the sum of the maximum lesion diameters was > 10 cm, 2 vials (1.0 × 10^12 vp) if the sum of the maximum lesion diameters was ≤ 10 cm. The cycle is 21 days up to 2-5 cycles.
  Arms: H101+Sorafenib
Drug: Sorafenib — Sorafenib will be administered as the original dose before enrollment, or be adjusted by the doctor according to the tolerance.

SUMMARY:
Sorafenib, as a first-line treatment for patients with advanced HCC, can significantly prolong the overall survival rate of patients. However, about 53-71% of patients showed stable disease (SD) after sorafenib treatment, and further studies to explore optimal therapy for these patients are still needed.

Oncolytic viruses are a type of virus that can selectively replicate in tumor cells and then destroy tumor cells, of which recombinant human adenovirus type 5 (H101) is the first oncolytic virus drug which was approved in the world. Recent studies indicate that H101 shows anti-tumor effects on liver cancer and there may be a synergistic effect between recombinant human adenovirus type 5 and sorafenib in the inhabitation of hepatoma cells in vitro. This study aims to further verify the effect and safety of recombinant human adenovirus type 5 combined with sorafenib in the treatment of advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
Primary liver cancer is the fourth most common malignant tumor and the second most lethal cause of tumor in China, mainly including Hepatocellular carcinoma (HCC) and Intrahepatic Cholangiocarcinoma. ICC) and HCC-ICC, among which hepatocellular carcinoma accounts for about 75% of all primary liver cancer, bringing a heavy disease burden to China's health system and society. At present, for patients with unresectable advanced liver cancer, the commonly used treatment options include transcatheter chemoembolization (TACE), systemic therapy and radiotherapy. Since the introduction of the molecular-targeted drug Sorafenib in 2007, a number of clinical studies have shown that sorafenib has benefits for patients with advanced liver cancer in different countries and regions and with different liver disease backgrounds. It has become the standard therapy for advanced HCC and has been recommended for first-line treatment of advanced HCC patients by guidelines of many countries. However, although sorafenib can significantly prolong the overall survival rate, about 53-71% of patients still show stable disease (SD) after treatment. For these patients, further exploration is needed to optimize the treatment.

Oncolytic viruses are a class of viruses that can selectively replicate in tumor cells and then lytic tumor cells. Among them, recombinant human adenovirus TYPE 5 H101 is the world's first commercially available oncolytic drug, which has been approved for the treatment of head and neck tumors in 2003. Recombinant human adenovirus type 5 (H101) is a kind of oncolytic adenovirus, which can selectively replicate in tumor cells with deficient tumor suppressor gene p53 by knocking out e1B-55KD gene and partial gene fragment (78.3 ~ 85.8μm) of E3 region of human adenovirus type 5. Based on the data from the head and neck tumor-related clinical trial of recombinant human adenovirus H101, the drug has been approved for the treatment of advanced nasopharyngeal carcinoma in China. Based the study found that in recent years, in addition to the head and neck cancer, human recombinant adenovirus type 5 H101 also displayed antitumor effect on liver cancer, and the selective killing effect of the low concentration H101 on liver cancer cell associated with p53 gene mutation, and the high concentration of H101 on liver cancer cell and immortalized the role of normal liver cells is not restricted by cell p53 status. In vitro studies showed that both H101 and sorafenib alone could significantly inhibit the proliferation and induce apoptosis of human hepatoma cell lines HepG2 and Hep3B, and the combined effect of the two drugs was more significant than that of single drug 16. The synergistic mechanism of recombinant adenovirus H101 and sorafenib may be related to the influence of Raf/MEK/ERK signaling pathway. Sorafenib can block Raf/MEK/ERK signal transduction pathway, thereby inhibiting angiogenesis, while down-regulating the expression level of anti-apoptotic protein McL-1, and further inducing apoptosis of tumor cells. Meanwhile, sorafenib can upregulate the expression of Coxsackie adenovirus receptor (CAR) on the surface of hepatocellular carcinoma cells, increase the sensitivity of tumor cells to adenovirus, and enhance the oncolytic effect of H101. In addition, H101 combined with sorafenib can also effectively inhibit the expression of VEGF, thereby inhibiting the proliferation of tumor cells.

Based on the human recombinant adenovirus type 5 show the joint sorafenib synergy and its potential for the curative effect of hepatocellular carcinoma, this research intends to carry out a prospectie, intrusive, single-arm study, further validation of human recombinant adenovirus type 5 joint sorafenib therapy efficacy and safety of primary liver cancer, provides evidence-based medical evidence to support for clinical medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years and ≤ 70 years of age, male or female
* Histologically/radiologically diagnosed advanced unresectable hepatocellular carcinoma
* Patients had received sorafenib as systemic therapy for advanced HCC with radiographic assessment of Stable Disease (SD) according to mRECIST criteria
* ECOG performance status of 0-2
* Child-Pugh score ≤ 7
* At least one measurable target lesion according to mRECIST and at least one lesion ≥ 10 mm; the lesions previously treated by radiotherapy or local regional therapy must have imaging evidence of disease progression to be considered as target lesions
* Life expectancy ≥ 3 months
* A) White blood cell count ≥ 3.0 × 10 ^ 9/L, absolute neutrophil count ≥ 3.0 × 10 ^ 9/L, platelet count ≥ 50 × 10 ^ 9/L, hemoglobin > 100 g/L; B) INR ≤ 1.5 times the upper limit of normal, APTT ≤ 1.5 times the upper limit of normal or PTT ≤ 1.5 times the upper limit of normal; C) Total bilirubin ≤ 2.5 times the upper limit of normal; ALT and AST ≤ 5 times the upper limit of normal; serum creatinine ≤ 1.5 times the upper limit of normal
* Voluntarily participate in this study and sign the informed consent
* Female patients of childbearing age or male patients with sexual partners of childbearing age should take effective contraceptive measures throughout the treatment period and 6 months after treatment

Exclusion Criteria:

* Pregnant or lactating women
* Diffuse liver cancer or tumor not amenable to mRECIST criteria
* Prior treatment with oncolytic virus (e.g., T-VEC)
* Patients who are known to be allergic to the study drug or its active ingredients
* Sorafenib administration < 14 days
* History of immunodeficiency or autoimmune disease, or chronic systemic steroid therapy or any form of immunosuppressive therapy within 7 days prior to enrollment
* Patients with any other unstable systemic disease or other malignancy that may reduce life expectancy
* Patients participate in another interventional clinical trial within 30 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-12-28 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) according to mRECIST criteria | From the first administration of the study drug to disease progression, occurrence of unacceptable toxicity, withdrawal of informed consent or termination of the study (assessed up to 24 months)
  MRECIST criteria are based on traditional RECIST V1.0 and combined with specific assessment of hepatocellular carcinoma (HCC) (active lesions vs. Necrosis/fibrous nodules) to evaluate the efficacy of HCC

SECONDARY OUTCOMES:
Changes from baseline in alpha-fetoprotein (AFP) serum levels | 1 year
  Alpha-fetoprotein (AFP) is a protein produced in the liver and also the most widely accepted serum biomarker used in the management of hepatocellular carcinoma (HCC). Monitoring the serum level of AFP may provide important prognostic value. The serum levels of AFP will be obtained at baseline before treatment and then monitored during treatment and follow-up (every six weeks) to evaluate the effect of investigated drugs.
Disease control rate (DCR) | From the first administration of the study drug to disease progression, occurrence of unacceptable toxicity, withdrawal of informed consent or termination of the study (up to 1 year)
  The disease control rate is the sum of complete response rate, partial response rate and disease stability rate, that is, the ratio of patients with complete response, partial response and disease stability to all assessable patients.
Progression-free survival (PFS) | up to 1 year
  The total length of time from the onset of treatment and the observation of disease progression or the occurrence of death from any cause
1 year survival rate | 1 year
  The proportion of patients who survive 1years or more with each combination of treatments.
Number of participants with adverse events | 1 year
  The number of patients who had a medical event during treatment that was not necessarily causally related to the drug used, according to CTCAE V5.0

CONTACTS AND LOCATIONS:
Overall Officials: Chang Liu, MD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (4):
- China (4):
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Tangdu Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi